CLINICAL TRIAL: NCT06830187
Title: Radiological and Audiological Correlation in Otosclerosis: a Prospective Case-Control Study Evaluating Temporal Bone CT, Bone Mineral Density, and Hearing Loss
Brief Title: Investigating the Relationship Between Temporal Bone CT, Bone Density, and Hearing Loss in Otosclerosis Patients
Status: Recruiting | Type: Observational
Sponsor: İbrahim Emir Yeşil (Other)
Responsible Party: Sponsor-Investigator, İbrahim Emir Yeşil, MD, Otorhinolaryngologist, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: HacettepeU-SBA 24/365
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Otosclerosis of Middle Ear; Bone Density; Vitamin D Deficiency
Keywords: Otosclerosis; Temporal Bone CT; Bone Mineral Density (BMD); Serum Vitamin D; Audiology; Stapedectomy; Hounsfield Units
MeSH Terms: conditions — Vitamin D Deficiency; Otosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Otosclerosis Group: Participants diagnosed with otosclerosis based on clinical and audiological criteria. These individuals have undergone or are planned for stapedectomy or stapedotomy surgery. High-resolution CT scans and bone metabolism markers will be analyzed to assess correlations with disease severity.
- Control Group: Individuals without otosclerosis who have undergone temporal bone CT imaging for unrelated reasons. They have no history of conductive or mixed hearing loss. Their imaging and metabolic parameters will be compared with those of the otosclerosis patients to identify significant differences.

SUMMARY:
The goal of this observational case-control study is to evaluate the relationship between temporal bone computed tomography (CT) findings, bone mineral density (BMD), and audiological parameters in adults diagnosed with otosclerosis. The main questions it aims to answer are:

Is there a correlation between temporal bone CT density values and the severity of hearing loss in otosclerosis? Do bone mineral density and serum vitamin D levels differ between otosclerosis patients and individuals without otosclerosis? Researchers will compare patients diagnosed with otosclerosis to a control group without otosclerosis to determine if CT-based density variations are associated with disease severity and systemic bone metabolism markers.

Participants who have already had a temporal bone CT scan as part of their routine clinical evaluation will undergo:

Bone mineral density (BMD) assessment via dual-energy X-ray absorptiometry (DEXA) Serum vitamin D level measurement Audiological testing, including pure tone audiometry and speech discrimination tests This study aims to improve the diagnostic and prognostic understanding of otosclerosis by integrating imaging, metabolic, and audiological data.

ELIGIBILITY:
Inclusion Criteria (Otosclerosis Group):

* Adults diagnosed with otosclerosis based on audiological and clinical assessment
* Patients with available high-resolution CT scans and audiological data
* Individuals who have undergone stapedectomy or stapedotomy surgery
* Availability of bone mineral density and serum vitamin D data

Inclusion Criteria (Control Group):

* Patients without otosclerosis but with temporal CT imaging for other indications
* No history of conductive or mixed hearing loss
* Availability of BMD and vitamin D data

Exclusion Criteria:

* History of primary metabolic bone diseases (osteoporosis, Paget's disease)
* Use of medications affecting bone metabolism (bisphosphonates, corticosteroids)
* History of chronic otitis media or prior ear surgeries
* Patients who received head and neck radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients evaluated at the Otorhinolaryngology Department of Hacettepe University for hearing-related concerns. Participants will be selected from individuals who have undergone audiological testing and temporal bone computed tomography (CT) imaging as part of their clinical assessment.
  The study includes two groups:
  Otosclerosis Patients (Study Group): Adults diagnosed with otosclerosis based on clinical, audiological, and radiological criteria. These patients have undergone or are scheduled for stapedectomy or stapedotomy surgery.
  Non-Otosclerosis Patients (Control Group): Individuals who have no clinical or audiological signs of otosclerosis but have undergone temporal bone CT for unrelated reasons, such as investigation of other otologic symptoms (e.g., vertigo, tinnitus, or trauma assessment).
  Participants will primarily be recruited from tertiary care settings within the hospital, ensuring access to specialized diagnostic and surgical inter
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Temporal Bone CT Density Measurements | Baseline (Preoperative assessment)
  Measurement of bone density at key anatomical sites including the stapes footplate, oval window, and otic capsule, using Hounsfield Units (HU) from high-resolution temporal bone CT scans.
Pure Tone Audiometry (PTA) Thresholds | Baseline (Preoperative assessment)
  Hearing thresholds will be assessed using pure tone audiometry (PTA) across standard frequencies (500 Hz, 1000 Hz, 2000 Hz, 4000 Hz). The average PTA threshold (in dB HL) will be reported to evaluate the severity of hearing impairment.
Air-Bone Gap (ABG) Measurement | Baseline (Preoperative assessment)
  Air-bone gap (ABG) will be assessed at key frequencies (500 Hz, 1000 Hz, 2000 Hz, 4000 Hz) using pure tone audiometry. The mean ABG value (in dB HL) will be reported to evaluate the degree of conductive hearing loss.
Bone Mineral Density (BMD) Scores | Baseline (Preoperative assessment)
  Measurement of bone mineral density in lumbar spine and femoral neck using Dual-Energy X-ray Absorptiometry (DEXA) to explore systemic bone metabolism in otosclerosis patients.
Serum Vitamin D Levels | Baseline (Preoperative assessment)
  Measurement of 25-hydroxyvitamin D levels in blood samples to assess vitamin D status and its potential correlation with otosclerosis progression.

SECONDARY OUTCOMES:
Correlation Between CT Density and Audiological Parameters | Baseline (Preoperative assessment)
  Analysis of the relationship between preoperative CT bone density values and audiometric findings to determine if CT markers predict hearing loss severity.
Association Between Otosclerosis Severity and BMD/Vitamin D Levels | Baseline (Preoperative assessment)
  Statistical analysis to determine whether systemic bone metabolism markers (BMD, serum vitamin D) correlate with otosclerosis severity, as assessed by CT and audiological tests.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Atay, Assoc Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University Hospitals, Ankara, Turkey (Türkiye)